CLINICAL TRIAL: NCT02977091
Title: Fitness Level in Short Stature Children and After Growth Hormone Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Dror Nitsan, M.D, Meir Medical Center
Other Study IDs: 0258-16-MMC
Record Dates: First submitted 2016-11-21; First posted 2016-11-30 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Fitness
Keywords: short stature; fitness; children
MeSH Terms: conditions — Dwarfism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- GH deficiency or idiopathic short stature: growth hormone (GH) deficiency or idiopathic short stature children before they start GH treatment
  Interventions: Other: change in fitness level
- short stature: healthy short children
  Interventions: Other: change in fitness level

INTERVENTIONS:
Other: change in fitness level — fitness level assessed by the Euro-fit tests for school age children.including 1.body fat 2. single leg balance test 3.Plate Tapping -for speed of limb movement 4.Sit-and-Reach flexibility test 5. Standing Broad Jump - measures explosive leg power. 6.Handgrip Test - measures static arm strength 7.Sit-Ups in 30 seconds - measures trunk strength 8.Bent Arm Hang - muscular endurance/functional strength 9.20 m endurance shuttle-run - cardiorespiratory endurance Wingate anaerobic test which is a 30 seconds maximum pedaling against resistance on bike for evaluating the anaerobic fitness

SUMMARY:
fitness and Physical activity will be evaluate in short stature children, using the Euro Fitness testing and the Wingate anaerobic test. the fitness level will be evaluate in healthy short children and with growth hormone deficiency at base line and after 6 month .

DETAILED DESCRIPTION:
The Euro Fitness testing which is a series of field testing for children evaluating aerobic, strength and flexibility and the Wingate anaerobic test which is a 30 seconds maximum pedaling against resistance on bike for evaluating the anaerobic fitness.

the fitness test will be done in healthy short stature children and in growth hormone deficiency or idiopathic short stature from the endocrine unit in Meir medical center The test will be done at base line and after 6 month . The fitness test in child with growth hormone deficiency will be done before starting GH treatment and 6 month later.

The child will be asked to fill a questioner about his daily physical activity Anthropometric measurement will be taking including weight, height and fat percent. Details about age, sex, tanner stage, indication for growth hormone, dose, insulin growth factor-1 (IGF1) level will be taken from the medical file.

ELIGIBILITY:
Inclusion Criteria:

* short stature
* Physical healthy
* Mental healthy
* Capable to perform fitness test

Exclusion Criteria:

* Cardiac disease that interfere or risk the child during physical activity
* Respiratory disease that interfere or risk the child during physical activity
* Musculoskeletal disease interfering physical preformance.
* Family history of death for unknown reasons at an early age.
* Uncontroled thyroid diseae

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: short stature children
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
change in fitness level | change of fitness levels from base line and after 6 month in short children

CONTACTS AND LOCATIONS:
Overall Officials: Nitsan Dror, MD, Principal Investigator — senior in pediatric medicine
Locations (1):
- Meir Medical Center endocrine unit, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bar-Or O. The Wingate anaerobic test. An update on methodology, reliability and validity. Sports Med. 1987 Nov-Dec;4(6):381-94. doi: 10.2165/00007256-198704060-00001. No abstract available. PMID 3324256
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Ranson R, Stratton G, Taylor SR. Digit ratio (2D:4D) and physical fitness (Eurofit test battery) in school children. Early Hum Dev. 2015 May;91(5):327-31. doi: 10.1016/j.earlhumdev.2015.03.005. Epub 2015 Apr 4. PMID 25846842
- See also: The Eurofit Physical Fitness Test Battery — http://www.topendsports.com/testing/children.htm